CLINICAL TRIAL: NCT06099847
Title: Sacral Transcutaneous Electrical Stimulation Efficacy in Chronic Pelvic Pain: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nalan Capan Bolukbas, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/1719
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: transcutaneous electrical stimulation; chronic pelvic pain; sacral; randomized clinical trial

STUDY DESIGN:
Intervention Model Description: We aim to compare sacral TENS in patients with chronic pelvic pain and compare it with sham stimulation therapy.
Who Masked: Participant
Masking Description: Only participants are blinded for the intervention. Care provider (physiotherapist), investigator (medical doctor, physiatrist) and outcomes assessor (medical doctor, physiatrist) are not blinded and they are know which intervention (TENS or sham stimulation) is provided to the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Pelvic Pain Patients with TENS (Experimental): 19 patients with chronic pelvic pain have been received sacral TENS intervention.
  Interventions: Device: Sacral TENS Stimulation
- Chronic Pelvic Pain Patients with Sham Stimulation (Sham Comparator): 19 patients with chronic pelvic pain have been received sham stimulation intervention.
  Interventions: Device: Sham TENS Stimulation

INTERVENTIONS:
Device: Sham TENS Stimulation — Sacral TENS device without appropriate electrical stimulation have been applied to directly the skin of sacral area.
  Arms: Chronic Pelvic Pain Patients with Sham Stimulation
Device: Sacral TENS Stimulation — Sacral TENS stimulation have been applied to directly the skin of sacral area.
  Arms: Chronic Pelvic Pain Patients with TENS

SUMMARY:
The goal of this interventional study is to test of efficacy of sacral Transcutaneous Electrical Stimulation (TENS) in patients with chronic pelvic pain.

The main questions it aims to answer are:

1. Is sacral transcutaneous electrical stimulation (TENS) effective to reduce/relief pain in patients with chronic pelvic pain?
2. Is the effect of TENS comparable to sham stimulation therapy in patients with chronic pelvic pain?

DETAILED DESCRIPTION:
Our study aiming to test the efficacy of sacral transcutaneous electrical stimulation (TENS) intervention in patients with chronic pelvic pain. We aim to test the efficacy and compare it with sham stimulation therapy in chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Female with chronic pelvic pain for ≥6 months
* 18-65 years old
* Visual Numeric Scale of Pain score ≥4/10
* Voluntarily participate to the study

Exclusion Criteria:

* Pregnancy
* Having severe medical and/or psychiatric disorder
* Malignancy
* Chronic infection
* Inflammatory musculoskeletal system disease
* Skin infection in sacral/pelvic area
* Having implanted neuromodulatory device (such as pacemaker or defibrillator)
* Refusing to participate the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Visual Numeric Scale of Pain | Baseline (Before Treatment), immediately After Treatment and 1 Month After Treatment
  Patients with Chronic Pelvic Pain assessed their pain levels before, right after and 1 month after treatment

SECONDARY OUTCOMES:
The Pelvic Pain Impact Questionnaire | Baseline (Before Treatment), immediately After Treatment and 1 Month After Treatment
  Patients with Chronic Pelvic Pain assessed pelvic pain impact before, right after and 1 month after treatment
Female Sexual Function Index | Baseline (Before Treatment), immediately After Treatment and 1 Month After Treatment
  Patients with Chronic Pelvic Pain assessed their sexual functions before, right after and 1 month after treatment
Patient Satisfaction Questionnaire | Immediately After Treatment and 1 Month After Treatment
  Patients with Chronic Pelvic Pain assessed their satisfaction levels right after and 1 month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nalan Capan Bolukbas, M.D., Study Director — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arik MI, Kiloatar H, Aslan B, Icelli M. The effect of TENS for pain relief in women with primary dysmenorrhea: A systematic review and meta-analysis. Explore (NY). 2022 Jan-Feb;18(1):108-113. doi: 10.1016/j.explore.2020.08.005. Epub 2020 Aug 29. PMID 32917532
- [Result] Tirlapur SA, Vlismas A, Ball E, Khan KS. Nerve stimulation for chronic pelvic pain and bladder pain syndrome: a systematic review. Acta Obstet Gynecol Scand. 2013 Aug;92(8):881-7. doi: 10.1111/aogs.12184. Epub 2013 Jun 22. PMID 23710833
- See also: Main Reference — https://pubmed.ncbi.nlm.nih.gov/23710833/